CLINICAL TRIAL: NCT02618369
Title: Magnetic Resonance-Guided High Intensity Focused Ultrasound for Pain Management of Osteoid Osteoma and Benign Bone Tumors in Children and Young Adults
Brief Title: MR-Guided High Intensity Focused Ultrasound for Pain Management Of Osteoid Osteoma & Benign Bone Tumors in Children and Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, James Drake, Neurosurgeon, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1000040583
Record Dates: First submitted 2015-11-23; First posted 2015-12-01 (Estimated); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Osteoid Osteoma; Benign Bone Tumor; Pain
Keywords: High Intensity Focused Ultrasound
MeSH Terms: conditions — Osteoma, Osteoid; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MR-HIFU treatment (Other): The interventional radiologist will locate the target lesion and mark the volume to be treated using MRI images.
  The operator starts the treatment and monitors the progress of the treatment with MR thermal and dose maps to ensure adherence to treatment plan.
  Interventions: Device: MR-Guided High Intensity Focused Ultrasound

INTERVENTIONS:
Device: MR-Guided High Intensity Focused Ultrasound — Target treatment of bone lesion using High Intensity Focused Ultrasound

SUMMARY:
The Philips Sonalleve HIFU system is expected to be efficacious in reducing pain scores in patients with painful osteoid osteoma and other benign bone tumors, and in reducing their pain medication usage. No serious adverse effects are expected to result from this treatment.

DETAILED DESCRIPTION:
The objective of this study is to determine if MR-guided high-intensity focused ultrasound (MR-HIFU) is safe and effective technique for alleviating the pain associated with osteoid osteoma and other benign bone tumors in paediatric patients and adults(up to age 40 yrs). This technique meant to be an alternative to the standard-of-care, radiofrequency and laser-based percutaneous ablation. Safety of the technique will be assessed through evaluating non-targeted heating using MRI based temperature mapping. and inspecting patients post treatment for skin burns or other signs of serious adverse events. Efficacy of the technique will be assessed by evaluating/recording patients observed pain, quality of life, and pain medication usage both before and up to 6 months following treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 5-40 years.
* Able to give informed consent and have parent or guardian give informed consent if applicable.
* Weight <140 kg (requirement to fit safely on top of the HIFU table and inside the MRI).
* Definitive radiographic & clinical presentation of osteoid osteoma or other benign tumor lesion(avoiding need for biopsy).
* Pain specifically at the site of interest target lesion.
* Pain score for target lesion >/= 4 (indicating at least moderate pain) or an age-appropriate pain scale.
* Target lesion is uncomplicated (i.e. no fracture/spinal cord compression/cauda equina syndrome/soft tissue component).
* MR-HIFU treatment date >/= 2 weeks from most recent surgical treatment of lesion.

Exclusion Criteria:

* Unable to characterize pain specifically at the site of interest (target lesion).
* Pregnant/nursing females.
* Target lesion is complicated (i.e. presence of one of fracture/spinal cord compression/cauda equina syndrome/soft tissue component).
* Target lesion < 1cm from neurovascular bundles/bowel/hollow viscera or regions of cartilage/ bone growth).
* Target lesion located in skull, spine (excluding sacrum, which is allowed) or sternum.
* Scar along proposed HIFU beam path.
* Orthopaedic implant along proposed HIFU beam path or at site of target tissue.
* Serious cardiovascular, neurological, renal or haematological chronic disease.
* Active infection.
* Contraindication to general anaesthetic or gadolinium MRI contrast agent.
* Requirement for general anesthesia for non-HIFU related MRI's.

Ages: 5 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2014-04; Primary Completion 2018-04 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Change in pain intensity scores from baseline related to the site treated target lesion. | 2, 7, 14, 30 and 90 days following treatment.
  As measured on the pain diaries before and at day 2, 7, 14, 30 and 90 days after treatment.

SECONDARY OUTCOMES:
Reduction in in pain medication usage (NSAIDS, Opioids). | 2, 7, 14, 30 and 90 days following treatment.
  As noted in pain diaries by patient before and day 2, 7. 14, 30 and 90 days after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: James M Drake, FRCSC, FACS, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No